CLINICAL TRIAL: NCT06630728
Title: Addiction Potential of Very Low Nicotine Filtered Little Cigars
Acronym: LOWFLC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Dharini Bhammar, Assistant Professor, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2024C0053
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Smoking (Tobacco) Addiction
MeSH Terms: conditions — Smoking; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Smoking session (Experimental): All participants will undergo three smoking sessions: one using their own usual brand cigar, one with a normal nicotine study cigar, and one with a reduced nicotine study cigar
  Interventions: Drug: Reduced Nicotine Content Cigars; Drug: Normal nicotine content cigar; Drug: Usual brand cigar

INTERVENTIONS:
Drug: Reduced Nicotine Content Cigars — Participants will smoke a very low nicotine content filtered little cigar containing 0.50mg nicotine per gram of tobacco
  Other Names: VLNFLC
Drug: Normal nicotine content cigar — Participants will smoke a normal nicotine content filtered little cigar containing 5.17mg nicotine per gram of tobacco
  Other Names: FLC
Drug: Usual brand cigar — Participants will smoke their usual brand filtered little cigar
  Other Names: UB

SUMMARY:
The goal of this clinical trial is to learn how reducing the nicotine content in filtered little cigars can affect the the use of these cigars and lung health in current adult filtered little cigar users. The main question[s] it aims to answer are:

Are puffing behaviors, appeal/satisfaction, craving suppression, pharmacokinetic effects, and demand similar between the regular cigars smoked by participants, normal nicotine study cigars and very low nicotine study cigars? Are health effects and toxicant exposure similar between the regular cigars smoked by participants, normal nicotine study cigars and very low nicotine study cigars?

Participants will attend three study visits at OSU. Each visit would last up to 4 hours. During visits, they will

* fill several surveys
* provide blood samples
* perform breathing tests
* complete smoking sessions using either their own cigars or the study cigars.

ELIGIBILITY:
Inclusion Criteria:

* Smokers: 1) self-reported regular current filtered little cigars, cigarillos, little cigars, or small cigars use for the past 3 months; regular use will be defined as >=8 cigars smoked per month based on data showing median cigarillo use is 7.5 times per month and median FLC use is 14 times per month 59. We will attempt to bring in heavier users if feasible during recruitment; or 2) Cigarette smokers (>=8d/month for at least 3 months) with either (i) co-use of filtered little cigars, cigarillos, little cigars, or small cigars (at least once in their lifetime) or (ii) answering "yes" to the question "If all cigarettes were taken off the market, would you consider switching to filtered little cigars?"
* willing to abstain from all tobacco and nicotine for at least 12 hours prior to lab sessions
* Willing to bring their own, preferred brand little cigars/ small cigars/ cigarillos/ filtered little cigars to smoke in the lab on the first study visit
* capable of and willing to provide written informed consent
* read and speak in English.

Exclusion Criteria:

* Self-reported significant current lung disease (e.g. asthma, COPD, cystic fibrosis, pulmonary fibrosis); exercise-induced asthma, seasonal allergies for which a patient takes inhalers are allowed
* History of diagnosis or treatment for lung cancer
* Self-reported serious or uncontrolled kidney disease, liver disease, metabolic disease (thyroid, diabetes)
* History of cardiac event or distress within the past 3 months
* Unstable or significant psychiatric conditions (past and stable conditions will be allowed)
* Substance use disorders besides nicotine addiction
* Regular use of other tobacco products besides cigarettes such as snuff, chewing tobacco, snus, e-cigarettes >10d per month
* Exclusive large or premium cigar users
* Use of blunts every time or most of the time
* Regular use of cannabis >10d per month
* Planning to quit in next 30 days or currently trying to quit or quit attempt in past 30 days
* Pregnant, delivery in past 12 weeks, breastfeeding, or planning to get pregnant
* Inability to perform tests or follow instructions during testing

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Drug self-administration- Puff topography- total puff volume | During session 65 minute puffing session
  Derived from puff topography, total puff volume indicates the total amount of smoke inhaled during the smoking session. Units: mL
Forced expiratory volume in 1 second | Change from 0 to 65 minutes
  Spirometry will be completed before and after a 65 min smoking session
Nicotine | Change from 0 to 5 minutes
  Plasma sample will be analyzed for nicotine to assess pharmacokinetics from before to 5 minutes after the smoking session
Nicotine | Change from 0 to 65 minutes
  Plasma sample will be analyzed for nicotine to assess pharmacokinetics from before to 65 minutes after the smoking session
Carbon monoxide boost | Change from 0 to 5 minutes
  Exhaled carbon monoxide (CO) will be measured for assessing CO boost as a measure of toxicity before and 5 minutes after the smoking session
Carbon monoxide boost | Change from 0 to 65 minutes
  Exhaled carbon monoxide (CO) will be measured for assessing CO boost as a measure of toxicity before and after the smoking session

SECONDARY OUTCOMES:
Functional residual capacity | Change from 0 to 65 minutes
  Functional residual capacity will be measured with plethysmography to assess dynamic hyperinflation after the smoking session
Airway resistance (R5) | Change from 0 to 65 minutes
  Impulse oscillometry will be used to measure total airway resistance before and after the smoking session
Airway resistance (R5-R20) | Change from 0 to 65 minutes
  Impulse oscillometry will be used to measure small airway resistance before and after the smoking session
Modified Cigarette Evaluation Scale | 65 minutes
  The 12-item modified Cigarette Evaluation Scale will provide subjective effects of smoking cigars on a 0-6-point Likert scale from "not at all" to "extremely". There are five subscales including smoking satisfaction, psychological reward, enjoyment of respiratory symptoms, craving reduction, and aversion
Questionnaire on Smoking Urges (Tiffany Drobes) | Change from 0 to 5 minutes
  Smoking urges/craving will be measured using the Tiffany-Drobes Questionnaire of Smoking Urges: Brief Form. This is a 10-item measure where participants rate smoking-related items (All I want right now is a cigarette) on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Similar to previous studies, we will collapse the items into two previously identified factors (Factor 1: strong desire and intention to smoke; Factor 2: anticipation of relief from withdrawal symptoms). Scores are calculated by summing the items and range from 5 to 35 with higher scores indicating greater craving to smoke
Questionnaire on Smoking Urges (Tiffany Drobes) | Change from 0 to 65 minutes
  Smoking urges/craving will be measured using the Tiffany-Drobes Questionnaire of Smoking Urges: Brief Form. This is a 10-item measure where participants rate smoking-related items (All I want right now is a cigarette) on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). Similar to previous studies, we will collapse the items into two previously identified factors (Factor 1: strong desire and intention to smoke; Factor 2: anticipation of relief from withdrawal symptoms). Scores are calculated by summing the items and range from 5 to 35 with higher scores indicating greater craving to smoke
Minnesota Nicotine Withdrawal Scale | Change from 0 to 5 minutes
  Nicotine withdrawal will be assessed using the empirically validated 15-item version of the Minnesota Nicotine Withdrawal Scale (MNWS). Items were rated on a 5-point scale from 0 (none) to 4 (severe). This measure assesses smoking craving, anger/irritability, anxiety, depressed mood, restlessness/difficulty concentrating, increased appetite, sleep problems, and somatic symptoms (nausea, constipation, sore throat, dizziness, coughing). MNWS is the sum of 7 items with scores ranging from 0 to 28 and MNWS Craving is a single item with scores ranging from 0 to 4, higher scores indicate a greater craving.
Minnesota Nicotine Withdrawal Scale | Change from 0 to 65 minutes
  Nicotine withdrawal will be assessed using the empirically validated 15-item version of the Minnesota Nicotine Withdrawal Scale (MNWS). Items were rated on a 5-point scale from 0 (none) to 4 (severe). This measure assesses smoking craving, anger/irritability, anxiety, depressed mood, restlessness/difficulty concentrating, increased appetite, sleep problems, and somatic symptoms (nausea, constipation, sore throat, dizziness, coughing). MNWS is the sum of 7 items with scores ranging from 0 to 28 and MNWS Craving is a single item with scores ranging from 0 to 4, higher scores indicate a greater craving.
Hypothetical purchase task | 65 minutes
  Hypothetical purchase task offers a measure of relative reinforcing efficacy. It will be completed after each smoking session. It assesses how many cigars a participant would smoke in a 24-hour period at various hypothetical price conditions and has been used to characterize addiction potential for reduced nicotine content cigars vs. normal nicotine content cigars vs. usual brand cigars. Data from the task leads to five demand indices (intensity or consumption with no cost constraint, price point at which consumption becomes sensitive to price, breakpoint is the price where FLCs are no longer purchased because of high price, largest cost that a participant is willing to incur to purchase FLCs, and elasticity as a measure of the overall sensitivity of FLC consumption to escalating price that measures how behaviors would change under the constraint of increased price).
Cross-price task | 65 minutes
  The Cross-Price Task will estimate the substitutability of the study cigars for the usual brand cigars. It will be completed after each study product smoking session. Participants will be asked how many study products and usual products they would consume when the price of the study product is fixed and the usual product prices escalate. To determine the extent to which each alternative product serves as a substitute for the study product, cross-price elasticities (CPE) will be calculated as the slope of the regression line (B1) fit to the log-transformed mean purchasing of each study product when offered at fixed prices (C) versus log-transformed usual product price (P): logC = B0 + B1logP. CPE for each study product compared to UB product > 0.2 indicates substitution, CPE < -0.2 indicates complementarity, and CPE between -0.2 and 0.2 indicates independence of the two products

CONTACTS AND LOCATIONS:
Overall Officials: Dharini M Bhammar, PhD, MBBS, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No